CLINICAL TRIAL: NCT04524689
Title: Open-label, Phase 2 Study of Tusamitamab Ravtansine (SAR408701) Combined With Pembrolizumab and Tusamitamab Ravtansine (SAR408701) Combined With Pembrolizumab and Platinum-based Chemotherapy With or Without Pemetrexed in Patients With CEACAM5 Positive Expression Advanced/Metastatic Non-squamous Non-small-cell Lung Cancer (NSQ NSCLC)
Brief Title: Tusamitamab Ravtansine (SAR408701) in Combination With Pembrolizumab and Tusamitamab Ravtansine (SAR408701) in Combination With Pembrolizumab and Platinum-based Chemotherapy With or Without Pemetrexed in Patients With NSQ NSCLC
Acronym: CARMEN-LC05
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision, the decision is not related to any safety concern.
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACT16146; U1111-1233-9798 (Registry Identifier: ICTRP); 2023-509115-84 (Registry Identifier: CTIS)
Record Dates: First submitted 2020-08-20; First posted 2020-08-24 (Actual); Results first posted 2025-03-17 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-09

CONDITIONS: Non-squamous Non-small-cell Lung Cancer (NSQ NSCLC)
MeSH Terms: interventions — tusamitamab ravtansine; pembrolizumab; Cisplatin; Carboplatin; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Tusamitamab ravtasine 150 mg/m^2 + Pembrolizumab (Experimental): Pembrolizumab dose will be administered intravenously prior to intravenous administration of tusamitamab ravtansine dose every 3 weeks.
  Interventions: Drug: SAR408701 (Tusamitamab ravtansine); Drug: Pembrolizumab
- Tusamitamab ravtasine 170 mg/m^2 + Pembrolizumab (Experimental): Pembrolizumab dose will be administered intravenously prior to intravenous administration of tusamitamab ravtansine dose every 3 weeks.
  Interventions: Drug: SAR408701 (Tusamitamab ravtansine); Drug: Pembrolizumab
- Tusamitamab ravtansine 150 mg/m^2 + Pembrolizumab + carboplatin or cisplatin (Experimental): Pembrolizumab dose will be administered intravenously prior to intravenous adminstration of tusamitamab ravtansine dose every 3 weeks. Carboplatin will be infused over 15 to 60 minutes immediately after tusamitamab ravtansine infusion on Day 1 and Q3W for the first 4 cycles. Cisplatin will be infused approximately 30 minutes after tusamitamab ravtansine infusion on Day 1 and Q3W for the first 4 cycles.
  Interventions: Drug: SAR408701 (Tusamitamab ravtansine); Drug: Pembrolizumab; Drug: Cisplatin; Drug: Carboplatin
- Tusamitamab ravtansine 170 mg/m^2 + Pembrolizumab + carboplatin or cisplatin (Experimental): Pembrolizumab dose will be administered intravenously prior to intravenous adminstration of tusamitamab ravtansine dose every 3 weeks. Carboplatin will be infused over 15 to 60 minutes immediately after tusamitamab ravtansine infusion on Day 1 and Q3W for the first 4 cycles. Cisplatin will be infused approximately 30 minutes after tusamitamab ravtansine infusion on Day 1 and Q3W for the first 4 cycles.
  Interventions: Drug: SAR408701 (Tusamitamab ravtansine); Drug: Pembrolizumab; Drug: Cisplatin; Drug: Carboplatin
- Tusamitamab ravtansine 150 mg/m^2 + Pembrolizumab + carboplatin or cisplatin + pemetrexed (Experimental): Pembrolizumab dose will be administered intravenously prior to intravenous adminstration of tusamitamab ravtansine dose every 3 weeks. Pemetrexed will be infused over 10 minutes after tusamitamab ravtansine infusion on Day 1 and then Q3W. Carboplatin will be infused over 15 to 60 minutes immediately after pemetrexed infusion on Day 1 and Q3W for the first 4 cycles. Cisplatin will be infused approximately 30 minutes after pemetrexed infusion after pemetrexed infusion on Day 1 and Q3W for the first 4 cycles.
  Interventions: Drug: SAR408701 (Tusamitamab ravtansine); Drug: Pembrolizumab; Drug: Cisplatin; Drug: Carboplatin; Drug: Pemetrexed
- Tusamitamab ravtansine 170 mg/m^2 + Pembrolizumab + carboplatin or cisplatin + pemetrexed (Experimental): Pembrolizumab dose will be administered intravenously prior to intravenous adminstration of tusamitamab ravtansine dose every 3 weeks. Pemetrexed will be infused over 10 minutes after tusamitamab ravtansine infusion on Day 1 and then Q3W. Carboplatin will be infused over 15 to 60 minutes immediately after pemetrexed infusion on Day 1 and Q3W for the first 4 cycles. Cisplatin will be infused approximately 30 minutes after pemetrexed infusion after pemetrexed infusion on Day 1 and Q3W for the first 4 cycles.
  Interventions: Drug: SAR408701 (Tusamitamab ravtansine); Drug: Pembrolizumab; Drug: Cisplatin; Drug: Carboplatin; Drug: Pemetrexed

INTERVENTIONS:
Drug: SAR408701 (Tusamitamab ravtansine) — Pharmaceutical form:Concentrate for solution for infusion Route of administration: Intravenous
  Other Names: Tusamitamab ravtansine
Drug: Pembrolizumab — Pharmaceutical form: Concentrate for solution for infusion Route of administration: Intravenous
  Other Names: Keytruda
Drug: Cisplatin — Pharmaceutical form: Lyophilized powder for reconstitution in solution Route of administration: Intravenous
  Arms: Tusamitamab ravtansine 150 mg/m^2 + Pembrolizumab + carboplatin or cisplatin; Tusamitamab ravtansine 150 mg/m^2 + Pembrolizumab + carboplatin or cisplatin + pemetrexed; Tusamitamab ravtansine 170 mg/m^2 + Pembrolizumab + carboplatin or cisplatin; Tusamitamab ravtansine 170 mg/m^2 + Pembrolizumab + carboplatin or cisplatin + pemetrexed
Drug: Carboplatin — Pharmaceutical form: Concentrate for solution for infusion Route of administration: Intravenous
  Arms: Tusamitamab ravtansine 150 mg/m^2 + Pembrolizumab + carboplatin or cisplatin; Tusamitamab ravtansine 150 mg/m^2 + Pembrolizumab + carboplatin or cisplatin + pemetrexed; Tusamitamab ravtansine 170 mg/m^2 + Pembrolizumab + carboplatin or cisplatin; Tusamitamab ravtansine 170 mg/m^2 + Pembrolizumab + carboplatin or cisplatin + pemetrexed
Drug: Pemetrexed — Pharmaceutical form: Concentrate for solution for infusion Route of administration: Intravenous
  Arms: Tusamitamab ravtansine 150 mg/m^2 + Pembrolizumab + carboplatin or cisplatin + pemetrexed; Tusamitamab ravtansine 170 mg/m^2 + Pembrolizumab + carboplatin or cisplatin + pemetrexed

SUMMARY:
Primary Objective:

* Safety run-in part: to assess the tolerability and to determine the recommended doses of tusamitamab ravtansine in combination with pembrolizumab and tusamitamab ravtansine in combination with pembrolizumab and platinum-based chemotherapy with or without pemetrexed to be tested in the expansion part of the study in the NSQ NSCLC population
* Expansion part (including participants treated at the recommended dose for expansion [RDE] from the Safety Run-in part): to assess the antitumor activity of several dose levels (DLs; if applicable) of tusamitamab ravtansine in combination with pembrolizumab and of several DLs of tusamitamab ravtansine in combination with pembrolizumab, platinum-based chemotherapy, and pemetrexed in the NSQ NSCLC population

Secondary Objectives:

* To assess the safety and tolerability of several DLs (if applicable) of tusamitamab ravtansine in combination with pembrolizumab and of 1 DL of tusamitamab ravtansine in combination with pembrolizumab and platinum-based chemotherapy, and of several DLs of tusamitamab ravtansine in combination with pembrolizumab, and platinum-based chemotherapy with pemetrexed in the NSQ NSCLC population
* To assess the antitumor activity of several DLs (if applicable) of tusamitamab ravtansine in combination with pembrolizumab and of 1 DL of tusamitamab ravtansine in combination with pembrolizumab and platinum-based chemotherapy, and of several DLs of tusamitamab ravtansine in combination with pembrolizumab, platinum-based chemotherapy, and pemetrexed in the NSQ NSCLC population
* To assess the durability of the response to treatment with several DLs (if applicable) of tusamitamab ravtansine in combination with pembrolizumab and of 1 DL of tusamitamab ravtansine in combination with pembrolizumab and platinum-based chemotherapy, and of several DLs of tusamitamab ravtansine in combination with pembrolizumab and platinum-based chemotherapy, and pemetrexed in the NSQ NSCLC population
* To assess the antitumor activity of tusamitamab ravtansine in combination with pembrolizumab and platinum-based chemotherapy in the NSQ NSCLC population
* To assess the pharmacokinetics (PK) of tusamitamab ravtansine, pembrolizumab, pemetrexed, cisplatin, and carboplatin, each when given in combination as a doublet (tusamitamab ravtansine + pembrolizumab) or a triplet (tusamitamab ravtansine + pembrolizumab + platinum-based chemotherapy) or a quadruplet (tusamitamab ravtansine + pembrolizumab + platinum-based chemotherapy + pemetrexed)
* To assess the immunogenicity of tusamitamab ravtansine in combination with pembrolizumab and tusamitamab ravtansine in combination with pembrolizumab and platinum based chemotherapy with or without pemetrexed

DETAILED DESCRIPTION:
The expected duration of study intervention for participants may vary, based on disease progression date; median expected duration of study per participant is estimated at 10 months (up to 1 month for screening, a median of 6 months for treatment, a median of 1 month for EOT, and follow-up visit 90 days after the last IMP administration).

ELIGIBILITY:
Inclusion criteria :

* Histologically- or cytologically-confirmed diagnosis of advanced or metastatic NSQ NSCLC with no EGFR sensitizing mutation or BRAF mutation or ALK/ROS alterations.
* No prior systemic chemotherapy for the treatment of the participant's advanced or metastatic disease (treatment with chemotherapy and/or radiation as part of neoadjuvant/adjuvant therapy is allowed as long as completed at least 6 months prior to diagnosis of advanced or metastatic disease).
* Expression of CEACAM5 as demonstrated prospectively by a centrally assessed Immunohistochemistry (IHC) assay of ≥2+ in intensity involving at least 1% of the tumor cell population in archival tumor sample (or if not available fresh biopsy sample).
* Measurable disease based on RECIST 1.1.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies
* Life expectancy of at least 3 months

Exclusion criteria:

* Medical condition requiring concomitant administration of a medication with a strong CYP3A inhibitor.
* Uncontrolled brain metastases and history of leptomeningeal disease.
* Significant concomitant illness, including any severe medical condition that, in the opinion of the investigator or Sponsor, would impair the patient's participation in the study or interpretation of the results.
* History within the last 3 years of an invasive malignancy other than the one treated in this study, with the exception of resected/ablated basal or squamous-cell carcinoma of the skin or carcinoma in situ of the cervix, or other local tumors considered cured by local treatment.
* History of known acquired immunodeficiency syndrome (AIDS) related illnesses or known HIV disease requiring antiretroviral treatment, or active hepatitis A, B, or C infection.
* History of active autoimmune disease that has required systemic treatment in the past 2 years.
* History of allogeneic tissue/solid organ transplantation.
* Active infection requiring IV systemic therapy within 2 weeks prior to randomization or active tuberculosis.
* Interstitial lung disease or history of pneumonitis that has required oral or IV steroids
* Non-resolution of any prior treatment-related toxicity to < Grade 2 according to NCI CTCAE V5.0, with the exception of alopecia, vitiligo, or active thyroiditis controlled with hormone replacement therapy.
* Unresolved corneal disorder or any previous corneal disorder considered by an ophthalmologist to predict higher risk of drug-induced keratopathy. The use of contact lenses is not permitted.
* Symptomatic herpes zoster within 3 months prior to screening.
* Significant allergies to humanized monoclonal antibodies.
* Clinically significant multiple or severe drug allergies, intolerance to topical corticosteroids, or severe post-treatment hypersensitivity reactions (including, but not limited to, erythema multiforme major, linear immunoglobulin A [IgA] dermatosis, toxic epidermal necrolysis, and exfoliative dermatitis).
* Concurrent treatment with any other anticancer therapy.
* Have received prior chemotherapy treatment for advanced/metastatic NSCLC.
* The patient is a candidate for a curative treatment with either surgical resection and/or chemoradiation
* Washout period before the first administration of study intervention of less than 3 weeks or less than 5 times the half-life, whichever is shorter, for any investigational treatment).
* Any prior therapy targeting CEACAM5.
* Any prior treatment with any other anti-PD-1, or PD-L1 or programmed death ligand 2 (PD-L2), anti-CD137, or anti-cytotoxic T-lymphocyte-associated antigen-4.
* Any prior maytansinoid treatment (DM1 or DM4 ADC).
* Is receiving systemic steroid therapy ≤3 days prior to the first dose of study therapy or receiving any other form of immunosuppressive medication. Daily steroid replacement therapy or any corticosteroid premedication if applicable are allowed.
* Any radiation therapy to lung >30 Gy within 6 months of first study intervention administration.
* Has received or will receive a live vaccine within 30 days prior to the first study intervention administration.
* Any major surgery within the preceding 3 weeks of the first study intervention administration.

Prior/concurrent clinical study experience

* Current participation in any other clinical study involving an investigational study treatment or any other type of medical research.
* Poor organ function

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2020-10-26 (Actual); Primary Completion 2024-03-12 (Actual); Study Completion 2024-12-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (22):
- KU Medical Center_Investigational Site Number :8400002, Westwood, Kansas, United States
- Centro Avancado de Oncologia CECAN - Liga Contra o Cancer Site Number : 0760004, Natal, Rio Grande do Norte, Brazil
- Chile (4):
  - Centro de Investigacion y Desarrollo Oncologico (CIDO) Hochstetter 599 of. 602-603-1001, Temuco_Investigational Site Number :1520005, Temuco, La Araucanía
  - ONCOCENTRO APYS Av. La Marina 1702, 2do piso, Viña del Mar_Investigational Site Number :1520003, Viña del Mar, Región de Valparaíso
  - Orlandi Oncologia General Salvo 159, Providencia_Investigational Site Number :1520002, Santiago
  - ICEGCLINIC Avenida Serafín Zamora 190 Torre B, piso 4. La Florida_Investigational Site Number :1520006, Santiago
- Czechia (2):
  - Fakultní nemocnice Olomouc Onkologická klinika I.P. Pavlova 6_Site Number :2030001, Olomouc
  - Nemocnice AGEL Ostrava - Vitkovice Plicní oddělení Zalužanského 2214/35_Site Number :2030002, Ostrava - Vitkovice
- France (4):
  - Institut Sainte-Catherine 250 Chemin de Baigne-Pieds_Investigational Site Number :2500005, Avignon
  - CHRU BREST 5 Avenue Foch_Investigational Site Number :2500003, Brest
  - Centre François Magendie Hôpital du Haut Lévèque Av.de Magellan_Investigational Site Number :2500001, Pessac
  - Pôle régional de Cancérologie 2 rue de la Milèterie BP 577_Investigational Site Number :2500004, Poitiers
- Hungary (2):
  - Országos Onkológiai Intézet Ráth György u. 7_Investigational Site Number :3480002, Budapest
  - Veszprém Megyei Tüdőgyógyintézet 049/2 Hrsz_Investigational Site Number :3480004, Farkasgyepü
- Israel (2):
  - Investigational Site Number : 3760001, Ramat Gan
  - Investigational Site Number : 3760002, Tel Aviv
- Spain (6):
  - Investigational Site Number : 7240005, A Coruña, A Coruña [La Coruña]
  - Investigational Site Number : 7240006, Badalona, Catalunya [Cataluña]
  - Investigational Site Number : 7240007, Oviedo, Principality of Asturias
  - Investigational Site Number : 7240002, Las Palmas
  - Investigational Site Number : 7240004, Madrid
  - Investigational Site Number : 7240001, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: ACT16146 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=25189&tenant=MT_SNY_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 22 centers in 8 countries. A total of 68 participants were screened from 26 October 2020 to 19 December 2023, of which 11 were screen failures. Screen failures were mainly due to not meeting the eligibility criteria. The study was terminated due to the discontinuation of the overall development of tusamitamab ravtansine by the Sponsor.
Pre-assignment Details: A total of 57 participants were enrolled in either Part A [doublet cohort (tusamitamab ravtansine + pembrolizumab)], Part B [triplet cohort (tusamitamab ravtansine + pembrolizumab + platinum-based chemotherapy i.e., cisplatin or carboplatin)] or Part C [quadruplet cohort (tusamitamab ravtansine + pembrolizumab + platinum-based chemotherapy + pemetrexed)] of the study per Investigator's choice.
Groups:
- Tusamitamab Ravtansine 150 mg/m^2 + Pembrolizumab: In Part A (doublet cohort), participants received tusamitamab ravtansine 150 milligram per square meter (mg/m^2) along with pembrolizumab 200 milligram (mg) via intravenous (IV) infusion on Day 1 and then every 3 weeks (Q3W) until confirmed disease progression, unacceptable toxicity, new anticancer therapy initiation, death, or the participant's or Investigator's decision to stop the treatment.
- Tusamitamab Ravtansine 170 mg/m^2 + Pembrolizumab: In Part A (doublet cohort), participants received tusamitamab ravtansine 170 mg/m^2 along with pembrolizumab 200 mg via IV infusion on Day 1 and then Q3W until confirmed disease progression, unacceptable toxicity, new anticancer therapy initiation, death, or the participant's or Investigator's decision to stop the treatment.
- Tusamitamab Ravtansine 150 mg/m^2 + Pembrolizumab + Cisplatin/Carboplatin: In Part B (triplet cohort), participants received tusamitamab ravtansine 150 mg/m^2 along with pembrolizumab 200 mg and either cisplatin 75 mg/m^2 or carboplatin area under the curve (AUC) 5 via IV infusion on Day 1 of the first 4 cycles (each cycle was 3 weeks), and then tusamitamab ravtansine 150 mg/m^2 along with pembrolizumab 200 mg via IV infusion on Day 1 of subsequent cycles until confirmed disease progression, unacceptable toxicity, new anticancer therapy initiation, death, or the participant's or Investigator's decision to stop the treatment.
- Tusamitamab Ravtansine 170 mg/m^2 + Pembrolizumab + Cisplatin/Carboplatin: In Part B (triplet cohort), participants received tusamitamab ravtansine 170 mg/m^2 along with pembrolizumab 200 mg and either cisplatin 75 mg/m^2 or carboplatin AUC 5 via IV infusion on Day 1 of the first 4 cycles (each cycle was 3 weeks), and then tusamitamab ravtansine 170 mg/m^2 along with pembrolizumab 200 mg via IV infusion on Day 1 of subsequent cycles until confirmed disease progression, unacceptable toxicity, new anticancer therapy initiation, death, or the participant's or Investigator's decision to stop the treatment.
- Tusamitamab Ravtansine 150 mg/m^2 + Pembrolizumab + Cisplatin/Carboplatin + Pemetrexed: In Part C (quadruplet cohort), participants received tusamitamab ravtansine 150 mg/m^2 along with pembrolizumab 200 mg, pemetrexed 500 mg/m^2, and either cisplatin 75 mg/m^2 or carboplatin AUC 5 via IV infusion on Day 1 of the first 4 cycles (each cycle was 3 weeks), and then tusamitamab ravtansine 150 mg/m^2 along with pembrolizumab 200 mg and pemetrexed 500 mg/m^2 via IV infusion on Day 1 of subsequent cycles until confirmed disease progression, unacceptable toxicity, new anticancer therapy initiation, death, or the participant's or Investigator's decision to stop the treatment.
- Tusamitamab Ravtansine 170 mg/m^2 + Pembrolizumab + Cisplatin/Carboplatin + Pemetrexed: In Part C (quadruplet cohort), participants received tusamitamab ravtansine 170 mg/m^2 along with pembrolizumab 200 mg, pemetrexed 500 mg/m^2, and either cisplatin 75 mg/m^2 or carboplatin AUC 5 via IV infusion on Day 1 of the first 4 cycles (each cycle was 3 weeks), and then tusamitamab ravtansine 170 mg/m^2 along with pembrolizumab 200 mg and pemetrexed 500 mg/m^2 via IV infusion on Day 1 of subsequent cycles until confirmed disease progression, unacceptable toxicity, new anticancer therapy initiation, death, or the participant's or Investigator's decision to stop the treatment.
Period: Overall Study
Arm/Group | Tusamitamab Ravtansine 150 mg/m^2 + Pembrolizumab | Tusamitamab Ravtansine 170 mg/m^2 + Pembrolizumab | Tusamitamab Ravtansine 150 mg/m^2 + Pembrolizumab + Cisplatin/Carboplatin | Tusamitamab Ravtansine 170 mg/m^2 + Pembrolizumab + Cisplatin/Carboplatin | Tusamitamab Ravtansine 150 mg/m^2 + Pembrolizumab + Cisplatin/Carboplatin + Pemetrexed | Tusamitamab Ravtansine 170 mg/m^2 + Pembrolizumab + Cisplatin/Carboplatin + Pemetrexed
Started | 23 | 2 | 6 | 1 | 22 | 3
Completed | 7 | 1 | 4 | 1 | 16 | 2
Not Completed | 16 | 1 | 2 | 0 | 6 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0 | 2 | 0
Not completed — Study terminated by Sponsor | 6 | 0 | 1 | 0 | 4 | 0
Not completed — Not related to Coronavirus disease 2019 | 9 | 0 | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All-treated population included all participants assigned to study treatment and who actually received at least 1 dose of study treatment.
Groups:
- Tusamitamab Ravtansine 150 mg/m^2 + Pembrolizumab: In Part A (doublet cohort), participants received tusamitamab ravtansine 150 mg/m^2 along with pembrolizumab 200 mg via IV infusion on Day 1 and then Q3W until confirmed disease progression, unacceptable toxicity, new anticancer therapy initiation, death, or the participant's or Investigator's decision to stop the treatment.
- Tusamitamab Ravtansine 150 mg/m^2 + Pembrolizumab + Cisplatin/Carboplatin: In Part B (triplet cohort), participants received tusamitamab ravtansine 150 mg/m^2 along with pembrolizumab 200 mg and either cisplatin 75 mg/m^2 or carboplatin AUC 5 via IV infusion on Day 1 of the first 4 cycles (each cycle was 3 weeks), and then tusamitamab ravtansine 150 mg/m^2 along with pembrolizumab 200 mg via IV infusion on Day 1 of subsequent cycles until confirmed disease progression, unacceptable toxicity, new anticancer therapy initiation, death, or the participant's or Investigator's decision to stop the treatment.
- Total: Total of all reporting groups
Arm/Group | Tusamitamab Ravtansine 150 mg/m^2 + Pembrolizumab | Tusamitamab Ravtansine 170 mg/m^2 + Pembrolizumab | Tusamitamab Ravtansine 150 mg/m^2 + Pembrolizumab + Cisplatin/Carboplatin | Tusamitamab Ravtansine 170 mg/m^2 + Pembrolizumab + Cisplatin/Carboplatin | Tusamitamab Ravtansine 150 mg/m^2 + Pembrolizumab + Cisplatin/Carboplatin + Pemetrexed | Tusamitamab Ravtansine 170 mg/m^2 + Pembrolizumab + Cisplatin/Carboplatin + Pemetrexed | Total
Number analyzed (Participants) | 23 | 2 | 6 | 1 | 22 | 3 | 57
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 10 | 0 | 3 | 0 | 9 | 2 | 24
  65 to 74 years | 9 | 2 | 1 | 1 | 12 | 1 | 26
  ≥ 75 years | 4 | 0 | 2 | 0 | 1 | 0 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 1 | 3 | 0 | 9 | 1 | 25
  Male | 12 | 1 | 3 | 1 | 13 | 2 | 32
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 20 | 2 | 4 | 1 | 13 | 3 | 43
  Multiple | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Not reported | 0 | 0 | 1 | 0 | 8 | 0 | 9
  Unknown | 2 | 0 | 1 | 0 | 1 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: All Cohorts: Number of Participants With Study Drug-Related Dose-Limiting Toxicities (DLTs)
Description: DLTs were defined as: a) Hematological abnormalities: grade 4 neutropenia for 7 or more consecutive days, grade 3 to 4 neutropenia complicated by fever (temperature ≥38.5 degree Celsius on more than 1 occasion) or microbiologically or radiographically documented infection, grade ≥3 thrombocytopenia associated with clinically significant bleeding requiring clinical intervention; b) Non-hematological abnormalities: grade 4 non-hematologic adverse event (AE), except AE symptoms related to the underlying disease as per the Investigator's judgment, grade ≥3 keratopathy. In addition, any other AE that the recruiting Investigators and sponsor deemed to be dose-limiting, regardless of its grade, was also considered as DLT.
Time Frame: Cycle 1 Day 1 up to Cycle 1 Day 21 (cycle duration=3 weeks)
Population: DLT-evaluable population included participants who received 1 cycle with at least 80% of the intended dose for each study treatment of the combination during the safety run-in at both doses of tusamitamab ravtansine in Part A (doublet cohort), Part B (triplet cohort) or Part C (quadruplet cohort).
Measure: Count of Participants; unit: Participants
Arm/Group | Tusamitamab Ravtansine 150 mg/m^2 + Pembrolizumab | Tusamitamab Ravtansine 170 mg/m^2 + Pembrolizumab | Tusamitamab Ravtansine 150 mg/m^2 + Pembrolizumab + Cisplatin/Carboplatin | Tusamitamab Ravtansine 170 mg/m^2 + Pembrolizumab + Cisplatin/Carboplatin | Tusamitamab Ravtansine 150 mg/m^2 + Pembrolizumab + Cisplatin/Carboplatin + Pemetrexed | Tusamitamab Ravtansine 170 mg/m^2 + Pembrolizumab + Cisplatin/Carboplatin + Pemetrexed
Number analyzed (Participants) | 21 | 2 | 5 | 1 | 21 | 3
Participants | 0 | 0 | 0 | 0 | 0 | 1

2. Primary Outcome: Doublet Cohort: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants with a confirmed complete response (CR) or partial response (PR) as best overall response (BOR) per response evaluation criteria in solid tumors (RECIST) version (v) 1.1. CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 millimeter (mm). PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Tumor assessments performed at baseline, then every 6 weeks for first 24 weeks, and every 9 weeks thereafter, approximately 158.4 weeks
Population: All-treated population included all participants assigned to study treatment and who actually received at least 1 dose of study treatment. Data is reported for Part A (doublet cohort) at both tusamitamab ravtansine doses.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tusamitamab Ravtansine 150 mg/m^2 + Pembrolizumab | Tusamitamab Ravtansine 170 mg/m^2 + Pembrolizumab
Number analyzed (Participants) | 23 | 2
percentage of participants | 47.8 [26.82 to 69.41] | 0 [0.00 to 84.19]

3. Primary Outcome: Quadruplet Cohort: Objective Response Rate
Description: ORR was defined as the percentage of participants with a confirmed CR or PR as per RECIST v1.1. CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Tumor assessments performed at baseline, then every 6 weeks for first 24 weeks, and every 9 weeks thereafter, approximately 139.9 weeks
Population: All-treated population included all participants assigned to study treatment and who actually received at least 1 dose of study treatment. Data is reported for Part C (quadruplet cohort) at both tusamitamab ravtansine doses.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tusamitamab Ravtansine 150 mg/m^2 + Pembrolizumab + Cisplatin/Carboplatin + Pemetrexed | Tusamitamab Ravtansine 170 mg/m^2 + Pembrolizumab + Cisplatin/Carboplatin + Pemetrexed
Number analyzed (Participants) | 22 | 3
percentage of participants | 59.1 [36.35 to 79.29] | 66.7 [9.43 to 99.16]

4. Secondary Outcome: All Cohorts: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs)
Description: An AE was defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. A serious AE was defined as any untoward medical occurrence that, at any dose resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent disability/incapacity or was a congenital anomaly/birth defect. A TEAE was defined as an AE that developed, worsened or became serious during the treatment-emergent period.
Time Frame: From first dose of study treatment (Day 1) up to 30 days post last dose of study treatment, approximately 162.4 weeks (doublet), 117 weeks (triplet), and 143.9 weeks (quadruplet)
Population: All-treated population included all participants assigned to study treatment and who actually received at least 1 dose of study treatment. Data is reported for Part A (doublet cohort), Part B (triplet cohort) and Part C (quadruplet cohort) at both tusamitamab ravtansine doses.
Measure: Count of Participants; unit: Participants
Arm/Group | Tusamitamab Ravtansine 150 mg/m^2 + Pembrolizumab | Tusamitamab Ravtansine 170 mg/m^2 + Pembrolizumab | Tusamitamab Ravtansine 150 mg/m^2 + Pembrolizumab + Cisplatin/Carboplatin | Tusamitamab Ravtansine 170 mg/m^2 + Pembrolizumab + Cisplatin/Carboplatin | Tusamitamab Ravtansine 150 mg/m^2 + Pembrolizumab + Cisplatin/Carboplatin + Pemetrexed | Tusamitamab Ravtansine 170 mg/m^2 + Pembrolizumab + Cisplatin/Carboplatin + Pemetrexed
Number analyzed (Participants) | 23 | 2 | 6 | 1 | 22 | 3
Participants
  Any TEAE | 23 | 2 | 6 | 1 | 22 | 3
  Any TESAE | 9 | 0 | 1 | 1 | 11 | 2

5. Secondary Outcome: Doublet and Quadruplet Cohorts: Progression-free Survival (PFS)
Description: PFS was defined as the time from the first study treatment administration to the date of the first documented progressive disease (PD) or death due to any cause, whichever came first. PD was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (including the baseline sum if that was the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. Appearance of 1 or more new lesions was also considered progression.
Time Frame: Tumor assessments performed at baseline, then every 6 weeks for first 24 weeks, and every 9 weeks thereafter, approximately 158.4 weeks (doublet) and 139.9 weeks (quadruplet)
Population: All-treated population included all participants assigned to study treatment and who actually received at least 1 dose of study treatment. Data is reported for Part A (doublet cohort) and Part C (quadruplet cohort) at both tusamitamab ravtansine doses.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tusamitamab Ravtansine 150 mg/m^2 + Pembrolizumab | Tusamitamab Ravtansine 170 mg/m^2 + Pembrolizumab | Tusamitamab Ravtansine 150 mg/m^2 + Pembrolizumab + Cisplatin/Carboplatin + Pemetrexed | Tusamitamab Ravtansine 170 mg/m^2 + Pembrolizumab + Cisplatin/Carboplatin + Pemetrexed
Number analyzed (Participants) | 23 | 2 | 22 | 3
months | 28.45 [4.107 to NA] — NA indicates that the upper limit of 95% confidence interval (CI) was not estimable due to insufficient number of participants with events. | NA [2.891 to NA] — NA indicates that the median and upper limit of 95% CI were not estimable due to insufficient number of participants with events. | 11.56 [5.520 to 15.869] | NA [5.388 to NA] — NA indicates that the median and upper limit of 95% CI were not estimable due to insufficient number of participants with events.

6. Secondary Outcome: All Cohorts: Disease Control Rate (DCR)
Description: DCR was defined as percentage of participants with a confirmed CR, confirmed PR or stable disease (SD) as BOR per RECIST v1.1. CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. SD was defined as neither sufficient shrinkage from the baseline study to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study. PD was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (including the baseline sum if that was the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. Appearance of 1 or more new lesions was also considered progression.
Time Frame: Tumor assessments performed at baseline, then every 6 weeks for first 24 weeks, and every 9 weeks thereafter, approximately 158.4 weeks (doublet), 113 weeks (triplet), and 139.9 weeks (quadruplet)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tusamitamab Ravtansine 150 mg/m^2 + Pembrolizumab | Tusamitamab Ravtansine 170 mg/m^2 + Pembrolizumab | Tusamitamab Ravtansine 150 mg/m^2 + Pembrolizumab + Cisplatin/Carboplatin | Tusamitamab Ravtansine 170 mg/m^2 + Pembrolizumab + Cisplatin/Carboplatin | Tusamitamab Ravtansine 150 mg/m^2 + Pembrolizumab + Cisplatin/Carboplatin + Pemetrexed | Tusamitamab Ravtansine 170 mg/m^2 + Pembrolizumab + Cisplatin/Carboplatin + Pemetrexed
Number analyzed (Participants) | 23 | 2 | 6 | 1 | 22 | 3
percentage of participants | 82.6 [61.22 to 95.05] | 100 [15.81 to 100.00] | 100 [54.07 to 100.00] | 100 [2.50 to 100.00] | 81.8 [59.72 to 94.81] | 100 [29.24 to 100.00]

7. Secondary Outcome: All Cohorts: Duration of Response (DOR)
Description: DOR was defined as the time from first documented evidence of CR or PR until PD determined per RECIST v1.1 or death from any cause, whichever occurred first. CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. PD was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (including the baseline sum if that was the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. Appearance of 1 or more new lesions was also considered progression.
Time Frame: as for outcome 6
Population: All-treated population included all participants assigned to study treatment and who actually received at least 1 dose of study treatment. Only participants with confirmed CR or PR as BOR were included in the analysis. Data is reported for Part A (doublet cohort), Part B (triplet cohort) and Part C (quadruplet cohort) at both tusamitamab ravtansine doses.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tusamitamab Ravtansine 150 mg/m^2 + Pembrolizumab | Tusamitamab Ravtansine 170 mg/m^2 + Pembrolizumab | Tusamitamab Ravtansine 150 mg/m^2 + Pembrolizumab + Cisplatin/Carboplatin | Tusamitamab Ravtansine 170 mg/m^2 + Pembrolizumab + Cisplatin/Carboplatin | Tusamitamab Ravtansine 150 mg/m^2 + Pembrolizumab + Cisplatin/Carboplatin + Pemetrexed | Tusamitamab Ravtansine 170 mg/m^2 + Pembrolizumab + Cisplatin/Carboplatin + Pemetrexed
Number analyzed (Participants) | 11 | 0 | 4 | 0 | 13 | 2
months | NA [7.688 to NA] — NA indicates that the median and upper limit of 95% CI were not estimable due to insufficient number of participants with events. |  | 10.45 [7.589 to NA] — NA indicates that the upper limit of 95% CI was not estimable due to insufficient number of participants with events. |  | 12.02 [8.345 to 19.220] | NA [4.074 to NA] — NA indicates that the median and upper limit of 95% CI were not estimable due to insufficient number of participants with events.

8. Secondary Outcome: Triplet Cohort: Objective Response Rate
Description: as for outcome 3
Time Frame: Tumor assessments performed at baseline, then every 6 weeks for first 24 weeks, and every 9 weeks thereafter, approximately 113 weeks
Population: All-treated population included all participants assigned to study treatment and who actually received at least 1 dose of study treatment. Data is reported for Part B (triplet cohort) at both tusamitamab ravtansine doses.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tusamitamab Ravtansine 150 mg/m^2 + Pembrolizumab + Cisplatin/Carboplatin | Tusamitamab Ravtansine 170 mg/m^2 + Pembrolizumab + Cisplatin/Carboplatin
Number analyzed (Participants) | 6 | 1
percentage of participants | 66.7 [22.28 to 95.67] | 0 [0.00 to 97.50]

9. Secondary Outcome: All Cohorts: Trough Concentration (Ctrough) of Tusamitamab Ravtansine
Description: Blood samples were collected for the measurement of tusamitamab ravtansine concentrations.
Time Frame: Pre-dose on Day 1 of Cycle 2 (cycle duration=3 weeks)
Population: PK population included all participants from the all-treated population with at least 1 post-baseline PK concentration with adequate documentation of dosing and sampling dates and times. Only those participants with data collected at the specified timepoint are reported. Data is reported for Part A (doublet cohort), Part B (triplet cohort) and Part C (quadruplet cohort) at both tusamitamab ravtansine doses.
Measure: Mean (Standard Deviation); unit: microgram per milliliter (mcg/mL)
Arm/Group | Tusamitamab Ravtansine 150 mg/m^2 + Pembrolizumab | Tusamitamab Ravtansine 170 mg/m^2 + Pembrolizumab | Tusamitamab Ravtansine 150 mg/m^2 + Pembrolizumab + Cisplatin/Carboplatin | Tusamitamab Ravtansine 170 mg/m^2 + Pembrolizumab + Cisplatin/Carboplatin | Tusamitamab Ravtansine 150 mg/m^2 + Pembrolizumab + Cisplatin/Carboplatin + Pemetrexed | Tusamitamab Ravtansine 170 mg/m^2 + Pembrolizumab + Cisplatin/Carboplatin + Pemetrexed
Number analyzed (Participants) | 16 | 2 | 4 | 1 | 17 | 2
microgram per milliliter (mcg/mL) | 8.0 (3.5) | 11.7 (1.5) | 7.6 (8.0) | 0.0 (NA) — NA indicates that the standard deviation was not estimable for only 1 participant. | 4.8 (2.7) | 7.6 (0.9)

10. Secondary Outcome: All Cohorts: Ctrough of Pembrolizumab
Description: Blood samples were collected for the measurement of pembrolizumab concentrations.
Time Frame: Pre-dose on Day 1 of Cycle 2 (cycle duration=3 weeks)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Tusamitamab Ravtansine 150 mg/m^2 + Pembrolizumab | Tusamitamab Ravtansine 170 mg/m^2 + Pembrolizumab | Tusamitamab Ravtansine 150 mg/m^2 + Pembrolizumab + Cisplatin/Carboplatin | Tusamitamab Ravtansine 170 mg/m^2 + Pembrolizumab + Cisplatin/Carboplatin | Tusamitamab Ravtansine 150 mg/m^2 + Pembrolizumab + Cisplatin/Carboplatin + Pemetrexed | Tusamitamab Ravtansine 170 mg/m^2 + Pembrolizumab + Cisplatin/Carboplatin + Pemetrexed
Number analyzed (Participants) | 3 | 2 | 4 | 1 | 17 | 2
mcg/mL | 14.0 (2.2) | 16.9 (4.8) | 13.4 (5.7) | 14.1 (NA) — NA indicates that the standard deviation was not estimable for only 1 participant. | 13.2 (4.2) | 10.3 (1.3)

11. Secondary Outcome: Quadruplet Cohort: Plasma Concentration of Pemetrexed
Description: Blood samples were collected for the measurement of pemetrexed concentrations.
Time Frame: 30 minutes post-dose on Day 1 of Cycle 1 (cycle duration=3 weeks)
Population: PK population included all participants from the all-treated population with at least 1 post-baseline PK concentration with adequate documentation of dosing and sampling dates and times. Only those participants with data collected at the specified timepoint are reported. Data is reported for Part C (quadruplet cohort) at both tusamitamab ravtansine doses.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Tusamitamab Ravtansine 150 mg/m^2 + Pembrolizumab + Cisplatin/Carboplatin + Pemetrexed | Tusamitamab Ravtansine 170 mg/m^2 + Pembrolizumab + Cisplatin/Carboplatin + Pemetrexed
Number analyzed (Participants) | 19 | 3
mcg/mL | 68.5 (80.8) | 53.6 (48.3)

12. Secondary Outcome: Triplet and Quadruplet Cohorts: Total Plasma Concentration Observed at the End of Infusion (Ceoi) of Cisplatin
Description: Blood samples were collected for the measurement of cisplatin concentrations.
Time Frame: At end of infusion on Day 1 of Cycle 1 (cycle duration=3 weeks)
Population: PK population included all participants from the all-treated population with at least 1 post-baseline PK concentration with adequate documentation of dosing and sampling dates and times. Only those participants with data collected at the specified timepoint are reported. Data is reported for Part B (triplet cohort) and Part C (quadruplet cohort) at both tusamitamab ravtansine doses.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Tusamitamab Ravtansine 150 mg/m^2 + Pembrolizumab + Cisplatin/Carboplatin | Tusamitamab Ravtansine 170 mg/m^2 + Pembrolizumab + Cisplatin/Carboplatin | Tusamitamab Ravtansine 150 mg/m^2 + Pembrolizumab + Cisplatin/Carboplatin + Pemetrexed | Tusamitamab Ravtansine 170 mg/m^2 + Pembrolizumab + Cisplatin/Carboplatin + Pemetrexed
Number analyzed (Participants) | 1 | 0 | 8 | 0
mcg/mL | 3.3 (NA) — NA indicates that the standard deviation was not estimable for only 1 participant. |  | 3.9 (1.0) |

13. Secondary Outcome: Triplet and Quadruplet Cohorts: Total Plasma Concentration Observed at the End of Infusion of Carboplatin
Description: Blood samples were collected for the measurement of carboplatin concentrations.
Time Frame: At end of infusion on Day 1 of Cycle 1 (cycle duration=3 weeks)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Tusamitamab Ravtansine 150 mg/m^2 + Pembrolizumab + Cisplatin/Carboplatin | Tusamitamab Ravtansine 170 mg/m^2 + Pembrolizumab + Cisplatin/Carboplatin | Tusamitamab Ravtansine 150 mg/m^2 + Pembrolizumab + Cisplatin/Carboplatin + Pemetrexed | Tusamitamab Ravtansine 170 mg/m^2 + Pembrolizumab + Cisplatin/Carboplatin + Pemetrexed
Number analyzed (Participants) | 4 | 1 | 10 | 2
mcg/mL | 33.4 (5.0) | 20.8 (NA) — NA indicates that the standard deviation was not estimable for only 1 participant. | 36.7 (17.4) | 29.7 (1.5)

14. Secondary Outcome: All Cohorts: Number of Participants With Treatment-emergent Anti-Therapeutic Antibodies (ATAs) Against Tusamitamab Ravtansine
Description: Blood samples were collected to assess the presence of treatment-emergent ATA against tusamitamab ravtansine. ATA incidence was defined as the number of participants found to have treatment-emergent ATA response during the study.
Time Frame: as for outcome 4
Population: ATA population included all participants from the all-treated population with at least 1 post-baseline ATA result (negative, positive, or inconclusive). Data is reported for Part A (doublet cohort), Part B (triplet cohort) and Part C (quadruplet cohort) at both tusamitamab ravtansine doses.
Measure: Count of Participants; unit: Participants
Arm/Group | Tusamitamab Ravtansine 150 mg/m^2 + Pembrolizumab | Tusamitamab Ravtansine 170 mg/m^2 + Pembrolizumab | Tusamitamab Ravtansine 150 mg/m^2 + Pembrolizumab + Cisplatin/Carboplatin | Tusamitamab Ravtansine 170 mg/m^2 + Pembrolizumab + Cisplatin/Carboplatin | Tusamitamab Ravtansine 150 mg/m^2 + Pembrolizumab + Cisplatin/Carboplatin + Pemetrexed | Tusamitamab Ravtansine 170 mg/m^2 + Pembrolizumab + Cisplatin/Carboplatin + Pemetrexed
Number analyzed (Participants) | 19 | 2 | 6 | 1 | 20 | 3
Participants | 9 | 1 | 3 | 0 | 8 | 2

ADVERSE EVENTS:
Time Frame: From first dose of study treatment (Day 1) up to 30 days post last dose of study treatment, approximately 162.4 weeks (doublet), 117 weeks (triplet), and 143.9 weeks (quadruplet). All-cause mortality was collected from first dose of study treatment (Day 1) up to end of the study visit, approximately 198 weeks.
Description: Analysis was performed on all-treated population.
Arm/Group | Tusamitamab Ravtansine 150 mg/m^2 + Pembrolizumab | Tusamitamab Ravtansine 170 mg/m^2 + Pembrolizumab | Tusamitamab Ravtansine 150 mg/m^2 + Pembrolizumab + Cisplatin/Carboplatin | Tusamitamab Ravtansine 170 mg/m^2 + Pembrolizumab + Cisplatin/Carboplatin | Tusamitamab Ravtansine 150 mg/m^2 + Pembrolizumab + Cisplatin/Carboplatin + Pemetrexed | Tusamitamab Ravtansine 170 mg/m^2 + Pembrolizumab + Cisplatin/Carboplatin + Pemetrexed
All-Cause Mortality (participants affected / at risk) | 5/23 | 0/2 | 2/6 | 1/1 | 11/22 | 0/3
Serious Adverse Events (participants affected / at risk) | 9/23 | 0/2 | 1/6 | 1/1 | 11/22 | 2/3
Other Adverse Events (participants affected / at risk) | 22/23 | 2/2 | 6/6 | 1/1 | 19/22 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tusamitamab Ravtansine 150 mg/m^2 + Pembrolizumab (N=23) | Tusamitamab Ravtansine 170 mg/m^2 + Pembrolizumab (N=2) | Tusamitamab Ravtansine 150 mg/m^2 + Pembrolizumab + Cisplatin/Carboplatin (N=6) | Tusamitamab Ravtansine 170 mg/m^2 + Pembrolizumab + Cisplatin/Carboplatin (N=1) | Tusamitamab Ravtansine 150 mg/m^2 + Pembrolizumab + Cisplatin/Carboplatin + Pemetrexed (N=22) | Tusamitamab Ravtansine 170 mg/m^2 + Pembrolizumab + Cisplatin/Carboplatin + Pemetrexed (N=3)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia Aspiration (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Septic Shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vascular Device Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metastases To Meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colitis Ulcerative (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Oesophageal Fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumoperitoneum (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic Cytolysis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immune-Mediated Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Disease Progression (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
General Physical Health Deterioration (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-Cardiac Chest Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sudden Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toxicity To Various Agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tusamitamab Ravtansine 150 mg/m^2 + Pembrolizumab (N=23) | Tusamitamab Ravtansine 170 mg/m^2 + Pembrolizumab (N=2) | Tusamitamab Ravtansine 150 mg/m^2 + Pembrolizumab + Cisplatin/Carboplatin (N=6) | Tusamitamab Ravtansine 170 mg/m^2 + Pembrolizumab + Cisplatin/Carboplatin (N=1) | Tusamitamab Ravtansine 150 mg/m^2 + Pembrolizumab + Cisplatin/Carboplatin + Pemetrexed (N=22) | Tusamitamab Ravtansine 170 mg/m^2 + Pembrolizumab + Cisplatin/Carboplatin + Pemetrexed (N=3)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Purulence (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (1) | 0 (0)
Respiratory Tract Infection Viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1)
Anaemia Megaloblastic (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Immune-Mediated Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 3 (4) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Depressed Mood (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
Dysaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Monoparesis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neuropathy Peripheral (Nervous system disorders) | 6 (7) | 0 (0) | 1 (2) | 0 (0) | 9 (12) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 0 (0)
Peripheral Sensory Neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Polyneuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1)
Conjunctivitis Allergic (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 0 (0)
Dry Eye (Eye disorders) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 4 (5) | 0 (0)
Keratitis (Eye disorders) | 10 (18) | 1 (2) | 1 (1) | 0 (0) | 4 (4) | 0 (0)
Keratopathy (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 1 (2)
Lacrimation Increased (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 0 (0)
Punctate Keratitis (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vision Blurred (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 5 (5) | 0 (0)
Visual Acuity Reduced (Eye disorders) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 2 (2) | 2 (2)
Visual Impairment (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Hyperaemia (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 4 (4) | 0 (0)
Hypertensive Crisis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Dry Throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 6 (6) | 0 (0)
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Malignant Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal Dryness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Sputum Discoloured (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 6 (9) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 0 (0) | 2 (4) | 0 (0) | 10 (11) | 1 (4)
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 11 (19) | 3 (3)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Tongue Blistering (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 9 (10) | 1 (1)
Dry Skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 1 (1) | 0 (0) | 6 (11) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 0 (0)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal Discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Nephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal Failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Vulvovaginal Pruritus (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 8 (8) | 0 (0) | 4 (8) | 0 (0) | 13 (19) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Device Related Thrombosis (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Mucosal Inflammation (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Non-Cardiac Chest Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Oedema Peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 6 (10) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 0 (0)
Aspartate Aminotransferase Increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Blood Creatinine Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Weight Decreased (Investigations) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Infusion Related Reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (4) | 0 (0)
Rib Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device Material Opacification (Product Issues) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was terminated due to the discontinuation of the overall development of tusamitamab ravtansine by the Sponsor and the enrollment of new participants in this study had been stopped on 21 December 2023.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2023-08-21): https://cdn.clinicaltrials.gov/large-docs/89/NCT04524689/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-09): https://cdn.clinicaltrials.gov/large-docs/89/NCT04524689/SAP_001.pdf